CLINICAL TRIAL: NCT00054704
Title: An Investigation of the Antidepressant Efficacy of an Antiglutamatergic Agent in Bipolar Depression
Brief Title: Riluzole to Treat Depression in Bipolar Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Placebo was better than active drug.
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 030092; 03-M-0092 (Other: NIH CNS IRB)
Record Dates: First submitted 2003-02-06; First posted 2003-02-07 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2017-01

CONDITIONS: Bipolar Disorder
Keywords: Riluzole; Neuroprotective; Open-Label Study; Glutamate Dysfunction; Bipolar Mood Disorder; Bipolar Disorder; Mood Disorder
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Riluzole (Experimental): Riluzole was dispensed either once or twice a day as 50 mg tablets. Riluzole dosing began at 50 mg twice per day by mouth and was increased on a weekly basis by 50 mg, as tolerated, to achieve a dose of 200 mg/day. Dose escalations continued until at least a 50% reduction in depression (MADRS) scores, intolerable side effects, or study completion. Dose was raised on a weekly basis by 50 mg until the dose of 200 mg was achieved unless precluded by an adverse event. If significant side effects occurred, titration was slowed and doses were reduced under double-blind conditions. The maximum permitted dose of riluzole was 200 mg/day. Those subjects not tolerating a dosage of 50 mg/day were removed from the study.
  Interventions: Drug: Riluzole
- Placebo (Placebo Comparator): Placebo pills resembling 50 mg riluzole tables were dispensed either once or twice a day. Dosing began at 50 mg twice per day by mouth and was increased on a weekly basis by 50 mg, as tolerated, to achieve a dose of 200 mg/day. Dose escalations continued until at least a 50% reduction in depression (MADRS) scores, intolerable side effects, or study completion. Dose was raised on a weekly basis by 50 mg until the dose of 200 mg was achieved unless precluded by an adverse event. If significant side effects occurred, titration was slowed and doses were reduced under double-blind conditions. The maximum permitted dose of riluzole was 200 mg/day. Those subjects not tolerating a dosage of 50 mg/day were removed from the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riluzole — Riluzole
  Other Names: Rilutek
  Arms: Riluzole
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study examines if Riluzole, FDA approved for ALS, will improve symptoms of depression in Bipolar Disorder.

Purpose: This study will examine the safety and effectiveness of riluzole (Rilutek trademark) for short-term treatment of depression symptoms, such as depressed mood, psychomotor retardation, and excessive sleeping in patients with bipolar disease. Riluzole is approved by the Food and Drug Administration (FDA) to treat amyotrophic lateral sclerosis (ALS, also known as Lou Gehrig's disease). Preliminary findings of a study using riluzole to treat acute depression in patients with unipolar depression indicate that it may have antidepressant properties in some patients.

Patients between 18 and 70 years of age with bipolar I or II disorder without psychosis may be eligible for this 8-week study. Candidates must be currently depressed, must have had at least one previous major depressive episode, and must have failed to improve with prior treatment with at least one antidepressant. They will be screened with a medical history, physical examination, electrocardiogram (EKG), blood and urine tests, and psychiatric evaluation. A blood or urine sample will be analyzed for illegal drugs. Women of childbearing potential will have a pregnancy test.

Participants will begin an 8-week course of treatment, starting with a placebo (a sugar pill formulated to look like the active drug) and, at some point, switching to riluzole. In addition to drug treatment, participants will undergo the following procedures:

Physical examination and electrocardiogram (EKG) at the beginning and end of the study;

Weekly check of vital signs (temperature, blood pressure and heart rate);

Weekly 1-hour interviews consisting of psychiatric and psychomotor rating scales to assess treatment response;

Weekly blood tests to measure blood levels of riluzole and evaluate drug side effects.

At the end of the study, participants' psychiatric status will be reassessed and appropriate long-term psychiatric treatment arranged.

Atendemos pacientes de habla hispana.

We enroll eligible participants locally and from around the country. Travel arrangements are provided and costs covered by the National Institute of Mental Health (NIMH). (Arrangements vary by distance and by specific study.) After completing the study participants receive short-term follow-up care while transitioning back to a provider.

DETAILED DESCRIPTION:
The treatments for acute unipolar depression have been extensively researched. However, despite the availability of a wide range of antidepressant drugs, clinical trials indicate that 30% to 40% of depressed patients fail to respond to first-line antidepressant treatment, despite adequate dosage, duration, and compliance. Very few studies have examined the efficacy of somatic treatments for the acute phase of bipolar depression. Thus, there is a clear need to develop novel and improved therapeutics for bipolar depression. Recent preclinical studies suggest that antidepressants may exert delayed indirect effects on the glutamatergic system. Clinical data suggests that lamotrigine an inhibitor of glutamate release and the N-methyl-D-aspartate (NMDA) antagonist ketamine may have antidepressant effects. Finally, our group recently found in two separate studies that the glutamate modulating agent riluzole was effective in treatment-resistant unipolar and bipolar depression (Zarate et al 2004). Together, these data suggest that the glutamatergic system may play a role in the pathophysiology and treatment of depression, and that agents, which more directly reduce glutamatergic neurotransmission, may represent a novel class of antidepressants.

In this study, we propose to extend our findings from open-label studies with riluzole in treatment-resistant depression by investigating its efficacy in a double-blind placebo-controlled study in bipolar depression.

Patients, ages 18 to 70 years with a diagnosis of bipolar disorder I or II current episode depressed (without psychotic features), will be randomized to double-blind treated to receive either riluzole (50-200 mg/day) or placebo for a period of 8 weeks. Acute efficacy will be determined by demonstrating a greater response rate using specified criteria.

Approximately 78 patients with acute bipolar depression will be enrolled in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male or female subjects, 18-70 years of age.

Female subjects of childbearing potential must be using a medically accepted means of contraception.

Each subject must have a level of understanding sufficient to agree to all required tests and examinations.

Each subject must understand the nature of the study and must sign an informed consent document.

Subjects must fulfill the criteria bipolar I or II disorder, current episode depressed without psychotic features as defined in the Diagnostic and Statistical Manual (DSM-IV) based on clinical assessment and confirmed by the Structured Clinical Interview for DSM (SCID-P).

Subjects must have an initial score at Visit 1 and Visit 2 of at least 20 on the MADRS.

Current duration of depressive episode should be at least 4 weeks.

Subjects must have experienced, in the opinion of the investigator, at least one previous major depressive episode as defined in DSM-IV (not including the current major depressive episode).

EXCLUSION CRITERIA:

Presence of psychotic features.

Female subjects who are either pregnant or nursing.

Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.

Subjects with uncorrected hypothyroidism or hyperthyroidism.

Clinically significant abnormal laboratory tests.

Current or past blood dyscrasia.

Documented history of hypersensitivity or intolerance to riluzole.

DSM-IV substance abuse or dependence within the past 90 days. No alcohol or recreational drug use will be permitted during the study.

Treatment with an injectable depot neuroleptic within less than one dosing interval between depot neuroleptic injections prior to visit 2.

Treatment with a reversible monoamine oxidase inhibitor (MAOI), guanethidine, or guanadrel within 1 week or with fluoxetine within 5 weeks prior to Visit 2.

Treatment with any other concomitant medication with primarily central nervous system (CNS) activity, other than specified in Appendix A.

Treatment with clozapine or electroconvulsive therapy (ECT) within 4 weeks prior to Visit 2.

Current diagnosis of schizophrenia or other psychotic disorder as defined in the DSM-IV.

Current Axis I Anxiety Disorder that is clinically significant.

Judged clinically to be at serious suicidal risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altamura CA, Mauri MC, Ferrara A, Moro AR, D'Andrea G, Zamberlan F. Plasma and platelet excitatory amino acids in psychiatric disorders. Am J Psychiatry. 1993 Nov;150(11):1731-3. doi: 10.1176/ajp.150.11.1731. PMID 8214185
- [Background] Auer DP, Putz B, Kraft E, Lipinski B, Schill J, Holsboer F. Reduced glutamate in the anterior cingulate cortex in depression: an in vivo proton magnetic resonance spectroscopy study. Biol Psychiatry. 2000 Feb 15;47(4):305-13. doi: 10.1016/s0006-3223(99)00159-6. PMID 10686265
- [Background] Bae HJ, Lee YS, Kang DW, Koo JS, Yoon BW, Roh JK. Neuroprotective effect of low dose riluzole in gerbil model of transient global ischemia. Neurosci Lett. 2000 Nov 10;294(1):29-32. doi: 10.1016/s0304-3940(00)01536-6. PMID 11044579
- [Derived] Hejazi NS, Farmer CA, Oppenheimer M, Falodun TB, Park LT, Duncan WC Jr, Zarate CA Jr. The relationship between the HDRS insomnia items and polysomnographic (PSG) measures in individuals with treatment-resistant depression. J Psychiatr Res. 2022 Apr;148:27-33. doi: 10.1016/j.jpsychires.2022.01.022. Epub 2022 Jan 11. PMID 35092868
- [Derived] Park LT, Lener MS, Hopkins M, Iadorola N, Machado-Vieira R, Ballard E, Nugent A, Zarate CA Jr. A Double-Blind, Placebo-Controlled, Pilot Study of Riluzole Monotherapy for Acute Bipolar Depression. J Clin Psychopharmacol. 2017 Jun;37(3):355-358. doi: 10.1097/JCP.0000000000000693. PMID 28338546

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Riluzole | Placebo
Started | 8 | 11
Completed | 3 | 6
Not Completed | 5 | 5
Not completed — Lack of Efficacy | 2 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants randomized.
Groups:
- Riluzole: Riluzole was dispensed either once or twice a day as 50 mg tablets. Riluzole dosing began at 50 mg twice per day by mouth and was increased on a weekly basis by 50 mg, as tolerated, to achieve a dose of 200 mg/day. Dose escalations continued until at least a 50% reduction in depression (MADRS) scores, intolerable side effects, or study completion. Dose was raised on a weekly basis by 50 mg until the dose of 200 mg was achieved unless precluded by an adverse event. If significant side effects occurred, titration was slowed and doses were reduced under double-blind conditions. The maximum permitted dose of riluzole was be 200 mg/day. Those subjects not tolerating a dosage of 50 mg/day were removed from the study.
- Placebo: Placebo pills resembling 50 mg riluzole tables were dispensed either once or twice a day. Dosing began at 50 mg twice per day by mouth and was increased on a weekly basis by 50 mg, as tolerated, to achieve a dose of 200 mg/day. Dose escalations continued until at least a 50% reduction in depression (MADRS) scores, intolerable side effects, or study completion. Dose was raised on a weekly basis by 50 mg until the dose of 200 mg was achieved unless precluded by an adverse event. If significant side effects occurred, titration was slowed and doses were reduced under double-blind conditions. The maximum permitted dose of riluzole was be 200 mg/day. Those subjects not tolerating a dosage of 50 mg/day were removed from the study.
- Total: Total of all reporting groups
Arm/Group | Riluzole | Placebo | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.29 (15.00) | 48.73 (11.29) | 48.08 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: Participants]
  United States | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a clinician-rated assessment of depression symptoms. Patients were rated weekly on 10 symptoms on a scale of 0 to 6 for each item, where 0 indicated no symptoms and 6 indicated the highest severity of that symptom. Total scores range from 0 to 60, where a moderate severity of depression would be present with a score of at least 20.
Time Frame: 8 weeks
Population: Data from all patients were included in the analysis, except for one riluzole patient with missing data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 8 | 11
Units on a scale | 29.551 (2.481) | 23.723 (1.916)
Statistical Analysis 1: Comparison: Riluzole vs Placebo; The primary intent of this study was to compare the efficacy of riluzole to placebo in the treatment of overall depressive symptomatology of bipolar disorder subjects who were acutely depressed. Data from 8 riluzole and 11 placebo participants were analyzed due to missing data for one riluzole patient; Test type: Superiority or Other; p = .086, Mixed Models Analysis — A linear mixed model included drug, visit and their interaction as fixed factors. Subject was a random factor. The test here is for the main effect of drug; Baseline score was a covariate. Restricted maximum likelihood estimates were used with a compound symmetry covariance structure; Mean Difference (Net) = -5.828, 95% CI 2-sided [-12.590 to 0.934], Standard Error of Mean 3.182

ADVERSE EVENTS:
Time Frame: Adverse event data was collected systematically on a weekly basis throughout the course of 8 weeks of study. An inventory of individual symptoms was used to evaluate adverse events on a scale from none to severe.
Arm/Group | Riluzole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 7/8 | 8/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole (N=8) | Placebo (N=11)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Gastrointestinal Problems (Gastrointestinal disorders) | 5 (5) | 1 (1)
Decreased libido (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Dizziness (General disorders) | 3 (3) | 0 (0)
Headache (General disorders) | 1 (1) | 2 (2)
Dry mouth (General disorders) | 1 (1) | 1 (1)
Muscle, joint, or bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Nasal and throat problems (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Sleep problems (General disorders) | 5 (5) | 4 (4)
Memory problems (General disorders) | 2 (2) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1)
Concentration difficulty (General disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 3 (3) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated due to results suggesting the active drug was leading to worse outcomes than placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No